CLINICAL TRIAL: NCT02085798
Title: Post-authorization, Observational Study to Assess the Evolution in the Normal Clinical Practise of Patients With Recent Diagnosis of Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML), Depending on the Time of Active Treatment Initiated
Brief Title: Health Outcomes of Recently Diagnosed Myelodysplastic Syndrome (MDS)/Chronic Myelomonocytic Leukemia (CMML) Patients Depending on Treatment Strategy (Wait and See, Support, Active Treatment)
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-CELGENE-SP-006
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Myelodysplastic Syndrome; Leukemia, Myelomonocytic, Chronic
Keywords: Leukemia, Myelomonocytic, Chronic, myelodysplastic syndrome, Prospective, Treatment strategy, epidemiologic data
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — Vision, Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Low or intermediate-1 risk MDS patients according to IPSS
  Interventions: Other: Either Wait and See, or Supportive Treatment, or Active Treatment at physician discretion
- Group 2: Intermediate-2 risk MDS patients according to IPSS
  Interventions: Other: Either Wait and See, or Supportive Treatment, or Active Treatment at physician discretion
- Group 3: Any risk CMML patients according to CPSS
  Interventions: Other: Either Wait and See, or Supportive Treatment, or Active Treatment at physician discretion

INTERVENTIONS:
Other: Either Wait and See, or Supportive Treatment, or Active Treatment at physician discretion — As described above

SUMMARY:
Post-authorisation observational study to assess the evolution in normal clinical practice of patients recently diagnosed with myelodysplastic syndrome (MDS) or chronic myelomonocytic leukaemia (CMML), depending on the moment when active treatment is initiated. Subjects will be recruited from approximately 50 haematology sites in Spain.

DETAILED DESCRIPTION:
Observational, prospective, post-authorisation multicentre study.

The study will include patients with a recent diagnosis (< 3 months) of MDS or CMML, receiving immediate active/support treatment or for whom an observation approach ("wait and see") is initially adopted, as per normal clinical practice in each participating site.

The minimum follow-up period of a participant patient will be 36 months from recruitment, until survival can be documented, differentiating between

1. Patients starting immediate active treatment: data will be collected every 3 months or every time an event arises during the active treatment phase. After the final dose of the initial treatment therapy, data collection will take place every 6 months during the post-treatment follow-up phase, regardless of the number of times the patient attends medical appointments, up to a minimum of 36 months' follow-up from the start of active treatment.
2. Patients for whom initial treatment strategy is support treatment or observation: a minimum follow-up period of 36 months will be established from the date of inclusion in the study, with data collection every 6 months or whenever an event occurs, regardless of the number of times the patient attends a medical appointment. The need for treatment for MDS (o CMML, where applicable) during this period will be considered an event, after which data will be collected every 3 months or each time an event occurs during the entire active treatment phase. After the final dose of the initial treatment therapy, data collection will take place every 6 months during the post-treatment follow-up phase, regardless of the number of times the patient attends medical appointments, up to a minimum of 36 months' follow-up from the start of active treatment.

Patients will be included consecutively, without the treatment prescription decisions affecting the decision to include the patient in the study. Indeed, in order to ensure the presence of patients with MDS of different prognoses and of patients with CMML, inclusion will be stratified into the following three cohorts, each of which will include patients receiving immediate treatment and those initially opting for observation/support:

* Group 1: Patients with low or intermediate-1 risk MDS as per the International Prognostic Scoring System (IPSS) 1.
* Group 2: Patients with intermediate-2 or high risk MDS as per IPSS.
* Group 3: Patients with any type of CMML as per the prognosis index CMML Prognostic Scoring System (CPSS) 2.

A total of 600 patients are expected to be recruited from 50 sites.

Primary objective:

To assess clinical evolution from the time of diagnosis in patients with MDS or CMML, within normal clinical practice.

The study will assess event free survival (EFS) depending on the therapeutic strategy initially adopted by the investigator after a diagnosis of MDS or CMML under normal clinical practice conditions.

EFS is defined as the period of time elapsed between diagnosis of the condition (MDS or CMML) and the appearance of one of the following events:

* Progression of the disease, or
* All-cause death, or
* Appearance of a clinically significant condition requiring a change in initial therapeutic strategy, or
* Appearance of an adverse event* requiring treatment to be suspended. *This applies to all patients included in the study, under active or support treatment.

Secondary objectives:

1. To describe the demographic, clinical (including MDS or CMML classification as per WHO 2008 (5, 19)), and analytical characteristics of patients recently diagnosed with MDS or CMML. Clinical characteristics include a health assessment as per the CIRS-G scale (Cumulative Illness Rating Scale for Geriatrics), the comorbidity rating for SMD (MDS-CI) by Della Porta and Malcovatti, 20 or other scale used across all participating sites in normal clinical practice, and the performance status of the patient as per ECOG scale.
2. To describe the therapeutic strategies initially applied for patients with MDS or CMML, based on clinical characteristics (specific cytogenetic alterations, adverse events, etc.), age, health status (CIRS-G scale), ECOG and IPSS (IPSS-R) or CPSS, in addition to the reasons for adopting different initial therapeutic strategies.
3. To analyse the response of MDS/CMML to treatment based on the IWG ( International Working Group) response criteria in myelodysplasia, modified in 2006.
4. To describe patient evolution based on time-dependent response parameters.

   * Time to Progression of the disease (TTP) as per the IWG response criteria modified in 2006.
   * Evolution to acute myeloblastic leukaemia (AML) (median time until transformation into AML).
   * To analyse progression free survival (PFS) from inclusion in the study until documented progression of MDS or CMML or death during follow-up.
   * Overall survival (OS) measured from the date of diagnosis of the disease until date of all-cause death, where applicable.
   * Assessment of overall response rate of dependence on red blood cell and platelet transfusions.
5. To document the tolerance profile (safety) of the treatment administered under normal clinical practice conditions.
6. To describe the use of healthcare resources relating to the initial therapeutic strategy for MDS or CMML in normal clinical practice, which can be financially measured, and to explore the possible differences both between the treat/do not treat option and the different therapeutic regimens administered.
7. To describe clinically significant events requiring a change in initial therapeutic strategy (counting for EFS, the primary objective of the study).

ELIGIBILITY:
Inclusion Criteria:

-1. Male or female subjects, aged 18 years or older. 2. Subjects with documented diagose of MDS or CMML within the last 3 months prior to entering the study and naive to treatment.

3. Signed informed consent.

Exclusion Criteria:

* 1. Subjects participating in an interventional clinical trial 2. Subjects who do not agree to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recently diagnosed (within the last 3 months prior to entering the study) of SMD or CMML, naïve to active treatment.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Up to a minimum of 36 months' follow-up from the start of active treatment
  Period of time elapsed between diagnosis of the condition (MDS or CMML) and the appearance of one of an event: Progression of the disease, death (all causes), clinically significant condition requiring a change in initial therapeutic strategy, adverse event requiring treatment discontinuation

SECONDARY OUTCOMES:
Health Assesment/performance Status | Approximately 3 years
  Changes from baseline to end of study as per CIRS-G scale, MDS-CI, ECOG
Response to active treatment | Up to end of treatment for each patient
  Response to active treatment up to progressions
Patient evolution based on time-dependent response parameters | Approximately 3 years
  Time to progression, time to evolution to AML (median time until transformation into AML), Progression Free Survival (from inclusion into the study to documented progression or death), Overall Survival (from diagnosis to death, all causes), Overall rate of dependence on red blood cells and platelet transfusion
Adverse Events | Approximately 3 years
  Safety profile description of treatment under normal clinical practice conditions
Patient Description | Baseline
  Demography, Clinical history of MDS or CMML, Blood test, Relevant comorbidities variables

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Rafel, RML Advocacy, Study Director — Celgene Spain; Regina Garcia, MD, Principal Investigator — Hospital Clínico Virgen de la Victoria, Málaga, Spain; David Valcárcel, MD, Principal Investigator — Hospital Vall d'Hebron, Barcelona, Spain
Locations (50):
- Spain (50):
  - Hospital Universitario Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Universitario La Ribera, Alzira, Alicante
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Complejo Hospitalrio La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital Punta de Europa, Algeciras, Cádiz
  - Hospital Universitario Donostia, San Sebastián, Guipuzcoa
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Getafe, Getafe, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de Antequera, Hospital de Antequera, Málaga
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - Complejo Hospitalario Torrecárdenas, Almería
  - Parc de Salut Mar- Hospital del Mar, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Duran Reynals, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitari de Girona Josep Trueta, Girona
  - Hospital Can Misses, Ibiza Town
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - CHU-Insular, Las Palmas de Gran Canaria
  - Hospital de León, León
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Santa Lucía, Murcia
  - Complejo Universitario Hospitalario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llàtzer, Palma de Mallorca
  - Complejo Hospitalrio Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Santa Bárbara, Soria
  - Hospital Clínico Universitario Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza